CLINICAL TRIAL: NCT05675605
Title: A Phase I/II Study of Oral TY-1091 in Adult Patients With Advanced Solid Tumors, Including RET-Fusion Non-Small Cell Lung Cancer, RET-Mutation Medullary Thyroid Cancer, and Other Tumors With RET Alterations
Brief Title: A Study of TY-1091 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYKM3604102
Record Dates: First submitted 2022-12-09; First posted 2023-01-09 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: RET-altered Non Small Cell Lung Cancer; Medullary Thyroid Cancer; RET-altered Papillary Thyroid Cancer; Neoplasms
MeSH Terms: conditions — Carcinoma, Medullary; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Multiple doses of TY-1091 for oral administration. Intervention: Drug: TY-1091
  Interventions: Drug: TY-1091
- Phase 2 Dose Expansion (Experimental): Multiple doses of TY-1091 for oral administration. Intervention: Drug: TY-1091
  Interventions: Drug: TY-1091

INTERVENTIONS:
Drug: TY-1091 — TY-1091(10mg,100mg) , once a day, oral administration Dose level is from 20mg to 800mg

SUMMARY:
This is a Phase 1/2, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antineoplastic activity of TY-1091 administered orally in participants with medullary thyroid cancer (MTC), RET-altered NSCLC and other RET-altered solid tumors.

DETAILED DESCRIPTION:
The study consists of 2 parts, a dose-escalation part (Phase 1) and an expansion part (Phase 2). Part1 will enroll participants with advanced non-resectable NSCLC, advanced non-resectable thyroid cancer and other advanced solid tumors that have progressed following standard systemic therapy, have not adequately responded to standard systemic therapy, or the participants must be intolerant to or the Investigator has determined that treatment with standard therapy is not appropriate, or there must be no accepted standard therapy for their disease. A multicenter, open-label design is adopted for part2. According to the obtained data of safety, tolerability, PK characteristics, and preliminary efficacy of TY-1091, one or two doses will be selected to conduct a dose expansion trial, which includes 3 cohorts with 20-40 subjects in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis during dose escalation (Phase 1) - Pathologically documented, definitively diagnosed non-resectable advanced solid tumor.

   All participants treated at doses > 50 mg per day must have MTC, or a RET-altered solid tumor per assessment of tumor tissue and/or blood
   * In the expansion stage phase (Phase 2) , patients should fulfill the following criteria at Screening Patients with histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC, MTC, or other solid tumors.

   Subject must have a documented RET gene fusion or mutation by a CLIA certified or equivalent testing. Next-generation sequencing (NGS), quantitative polymerase chain reaction (qPCR) test or fluorescence in situ hybridization (FISH) can be used to determine molecular eligibility At least one measurable lesion as defined by RECIST 1.1, not previously irradiated and not chosen for biopsy during the screening period. Patients without RECIST 1.1 measurable disease will be eligible for enrollment in Cohort 5.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 with no sudden deterioration 2 weeks prior to the first dose of study treatment.
3. Life expectancy of at least 3 months.
4. Adequate organ functions.
5. Ability to swallow capsules and willing and able to provide written informed consent approved by institutional review board (IRB) or independent ethics committee (IEC).
6. Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and 6 months following the last dose of study treatment; this may include barrier methods such as condom or diaphragm with spermicidal gel.

Exclusion Criteria:

1. For NSCLC patients, a targetable mutation in EGFR or MET, targetable rearrangement involving ALK, ROS1 or NTRK1-3.
2. History of other previous cancer (except for squamous cell or basal-cell carcinoma of the skin, or any in situ carcinoma that has been completely resected), requiring therapy within the previous 5 years.
3. For MTC patients, clinically significant involvement in the trachea, esophagus or complete encasement of great vessels (e.g., aorta or pulmonary artery) that in the opinion of the Investigator, could result in life-threatening complications due to rapid tumor regression.
4. Symptomatic primary central nervous system (CNS) tumor or metastases; symptomatic leptomeningeal carcinomatosis; untreated spinal cord compression.
5. Cardiovascular and cerebrovascular diseases/symptoms/indications meeting any of the following conditions:

   Mean resting corrected QT interval (electrocardiogram interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTcF) ≥470 msec obtained from 3 electrocardiograms; Any clinically significant resting ECG abnormalities in rhythm, conduction, or morphology, such as complete left bundle branch block, second and third degree heart block, PR interval > 250 ms; Any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death in a first-degree relative under 40 years of age, or any concomitant medication known to prolong QT interval; Left ventricular ejection fraction (LVEF) < 50%; Patients with a previous history of decreased myocardial contractility who experienced relevant symptoms within 6 months prior to study drug administration: such as chronic congestive heart failure, pulmonary edema or decreased cardiac ejection fraction; Patients with a history of acute or chronic cardiovascular and cerebrovascular diseases who had relevant symptoms within 6 months prior to study drug administration: such as myocardial infarction, severe or unstable angina, cerebral infarction, cerebral hemorrhage or transient ischemic attack.
6. Patients who have received treatment within 14 days prior to the first dose or need to continue treatment with strong CYP3A4 inducers/strong inhibitors, CYP3A4/CYP2C9/CYP2C19 sensitive substrate with a narrow treatment window or strong p-glycoprotein inhibitors.
7. Systemic anti-tumor treatment such as standard chemotherapy, biological therapy and immunological drug therapy within 28 days prior to the first dose; targeted therapy within 14 days or 5 half-lives of the first dose (calculated as a long time); anti-tumor traditional Chinese traditional medicine treatment within 7 days prior to the first dose.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
(Phase 1 )Dose Limiting Toxicity (DLT) | First 25 days of dosing
(Phase 1) Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 12 months
(Phase 2) Overall Response Rate (ORR) | up to 24 weeks

SECONDARY OUTCOMES:
(Phase 1) Overall Response Rate (ORR) | up to 24 weeks
iORR | up to 24 weeks
DCR | up to 24 weeks
CBR | 1 year
DOR | Approximately 1 year
PFS | Up to approximately 33 months
OS | Up to approximately 33 months
(Phase 1 and 2) Pharmacokinetic Parameters Including Maximum Plasma Drug Concentration (Cmax) | First 46 days of dosing
(Phase 1 and 2) Pharmacokinetic Parameters Including Terminal Elimination Half-life (t1/2) | First 46 days of dosing
(Phase 1 ) AUC0-24 | First 46 days of dosing
(Phase 1 and 2) Pharmacokinetic Parameters Including Tmax | First 46 days of dosing
(Phase 1 and 2) Pharmacokinetic Parameters Including Cmin | First 46 days of dosing
(Phase 1 ) AUC0-t | First 46 days of dosing
(Phase 1 ) AUCinf | First 46 days of dosing
(Phase 1 ) inflearance rate constant (Kel) | First 46 days of dosing
(Phase 1 ) apparent clearance (CL/F) | First 46 days of dosing
(Phase 1 ) Vd/F | First 46 days of dosing
(Phase 1 ) mean residence time (MRTinf) | First 46 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Province Cancer Hosipital Cheng, Bachelor, Principal Investigator — Jilin Province Cancer Hospital
Locations (1):
- Jinlin Province Cancer Hosipital, Changchun, Jilin, China